CLINICAL TRIAL: NCT01620736
Title: Phase II Trial to Assess Effect of Raltegravir on HTLV-1 Proviral Load
Brief Title: Trial to Assess Effect of Raltegravir on HTLV-1 Proviral Load
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The clinical trial did not receive any funding.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WashU201109171
Record Dates: First submitted 2012-01-25; First posted 2012-06-15 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Human T-cell Leukemia Virus Type 1 Infection
Keywords: Raltegravir; HTLV; Integrase
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir (Experimental): Treatment with raltegravir for 8 wks
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg po bid

SUMMARY:
This is a study of the effect of raltegravir on human T-cell leukemia virus type 1 (HTLV-1) viral load in asymptomatic patients. The study will enroll 14 subjects for a period of 2 months of treatment and 1 month of followup. The study will assess the effect of raltegravir on virus load in peripheral blood lymphocytes, level of virus gene expression, and sites of viral integration.

DETAILED DESCRIPTION:
About 5% of HTLV-1 infected individuals develop lymphoma or myelopathy. High levels of virus replication are predictive of disease development. HTLV-1 exhibits lower levels of variation than HIV-1, suggesting that drug resistance is less likely to occur. Raltegravir was shown to inhibit HTLV-1 integration and replication in culture using concentrations achievable with the approved dose used in HIV-1 infected patients. Currently, no treatment is recommended for asymptomatic infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HTLV-1 infection: documentation may be serologic assay (ELISA, Western blot) and confirmed to be HTLV-1 rather than HTLV-2 by differential Western blot (e.g. Genelabs Diagnostics HTLV Blot 2.4) or PCR.
2. Adequate hematologic function within 14 days before enrollment: ANC > 1000 cells/mm3, platelet count > 75,000 cells/mm3.
3. Adequate hepatic function, transaminase < 3 times the upper limit of normal; bilirubin < 2.0.
4. Creatinine < 2.0
5. Karnofsky Performance Status at least 70
6. Age at least 18.
7. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
8. Female patients of child bearing potential must have a negative pregnancy test within 72 hrs of initiation of therapy. Female patients are either post-menopausal or surgically sterilized or willing to use two acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study. Male patients must agree to use two acceptable methods for contraception for the duration of the study. Women must avoid pregnancy and men avoid fathering children while in the study.
9. Inclusion of Women and Minorities: Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Acute active infection requiring therapy. Chronic therapy with potentially myelosuppressive agents is allowed provided that entry hematologic criteria are met.
2. Women who are pregnant or breastfeeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
3. Patient has received other investigational drugs with 14 days before enrollment
4. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Effects of raltegravir on HTLV-1 provirus load in asymptomatic individuals | 8 wks
  Measured by DNA PCR from peripheral blood mononuclear cell DNA at days 0, 1, 8, 15, 29, 43, and 56.

SECONDARY OUTCOMES:
Effects of raltegravir on proviral load in CD4+CD25+, CD4+CD25-, and CD8+ cell populations | 8 wks
  Measured by real time PCR with DNA from sorted peripheral blood mononuclear cell DNA at days 1, 8, 15, 29, 43, and 56.
Effects of raltegravir on number of LTR circles and level of proviral RNA expression in PBMCs | 8 wks
  1. Number of LTR circles measure by real time PCR on peripheral blood mononculear cell DNA at days 0, 1, 8, 15, 29, 43, and 56
  2. Level of Proviral RNA Expression in PBMCs measured by real time RT PCR on peripheral blood mononculear cell RNA at days 0, 1, 8, 15, 29, 43, and 56
Effects of raltegravir on viral integrase gene or other viral sequence changes | 8 wks
  Measured by automated sequence analysis of PCR amplified viral DNA obtained at days 0, 1, 8, 15, 29, 43, and 56
Effect of raltegravir on viral integration sites | 8 wks
  Measured by automated DNA analysis of oligonucleotide linked PCR amplified DNA from peripheral blood mononuclear cell DNA obtianed at days 0, 1, 8, 15, 29, 43,and 56
Tolerance of raltegravir in HTLV-1 infected individuals | 8 wks
  Assessed by physical exam, CBC, and serum chemistries on days 29 and 57 and

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, MD PhD, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Seegulam ME, Ratner L. Integrase inhibitors effective against human T-cell leukemia virus type 1. Antimicrob Agents Chemother. 2011 May;55(5):2011-7. doi: 10.1128/AAC.01413-10. Epub 2011 Feb 22. PMID 21343468